CLINICAL TRIAL: NCT02068001
Title: Changes in Food Preference and Food Cue Responsivity After Bariatric Surgery
Acronym: Verrukkelijk
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wageningen University (Other)
Collaborators: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NL45837.081.13
Record Dates: First submitted 2014-02-05; First posted 2014-02-20 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Roux-en-Y Gastric Bypass
MeSH Terms: interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RYGB: Food preference assessment in 100 patients at different timepoints, in a subset of 30 participants, also brain reward response to food cues will be assessed.
  Interventions: Procedure: Roux-en-Y Gastric Bypass

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass

SUMMARY:
It has been suggested that obese people are more sensitive to sensory and rewarding effects of food, aspects that mediate food preferences and intake. Individuals that underwent Roux-en-Y gastric bypass surgery frequently report changes in food preference. They indicate a decreased preference for highly rewarding energy dense foods. Changes in food preference might be related to alterations in central (brain) mechanisms, related to reward sensing. The smell and sight of food can be considered as anticipatory cues for the rewarding effects of food intake. The aim of this study is to determine the effect of gastric bypass surgery on (alterations in) food preferences. Secondly, this study aims at assessing the effect of gastric bypass surgery on the brain reward response when exposed to sight and smell of food stimuli with different sugar and fat contents.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for Roux-en-Y Gastric Bypass Surgery at Rijnstate hospital

Exclusion Criteria:

* Lack of appetite
* Having difficulties swallowing/eating
* Being a vegetarian
* Allergic to food product used as stimuli in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Morbidly obese individuals (age 18-55 years) scheduled for Roux-en-Y gastric bypass surgery at Rijnstate hospital, Arnhem
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Development of food preferences after Roux-en-Y gastric bypass surgery | Participants will be followed for two years after they undergo surgery
  Food preferences will be assessed 2 weeks before Roux-en-Y Gastric Bypass surgery and 2 months, 1 year and 2 years after surgery.
Change in brain reward response to food cues | Before and 2 months after surgery
  Two weeks before and two months after Roux-en-Y Gastric Bypass the brain reward response to the sight and smell of food will be assessed in a subset of 30 participants.

SECONDARY OUTCOMES:
Plasma levels of endocannabinoids and satiety hormones | Before and 2 months after surgery
  Two weeks before and two months after Roux-en-Y gastric bypass surgery, fasted plasma levels of endocannabinoids, ghrelin, leptin, adiponectin and Glucagon-Like Peptide will be assessed in a subset of 30 participants.

OTHER OUTCOMES:
Descriptives | Before surgery
  General subject characteristics, e.g. age, gender, restrained eating score and other lifestyle and medical parameters.
  For the subset of 30 patients that participate in the fMRI measurements: disinhibition scores will be assessed.
Appetite ratings | During fMRI measurements, i.e., before and two months after surgery
  In a subset of 30 participants.
Olfactory performance | At each fMRI measurement, i.e., before and two months after surgery
  The Sniffin' Sticks test will be used to assess olfactory performance in the subset of 30 participants that will participate in the fMRI measurements. The sum-score of threshold, discrimination and identification tests will be used to determine if a participant is normosmic. A score of > 30 indicates a participant is normosmic.
Development of BMI | Before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne EM de Bruijn, MSc, Principal Investigator — Wageningen University; Harriët FA Zoon, MSc, Principal Investigator — Wageningen University
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem, Gelderland
  - Gelderse Vallei Hospital, Ede, Gelderland
  - Wageningen University, Wageningen, Gelderland